CLINICAL TRIAL: NCT05465408
Title: Addressing Non-Initiation of Recommended Adjuvant Endocrine Therapy With a Culturally Informed-Intervention
Brief Title: Culturally Aware AET Non-Initiation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jamie Jacobs, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-091
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Survivorship; Treatment Compliance; Treatment Adherence; Treatment Refusal
Keywords: Breast Cancer; Survivors; Hormone Therapy; Treatment Refusal; Treatment Compliance; Treatment Adherence
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance; Treatment Adherence and Compliance; Treatment Refusal | interventions — beta-Aminoethyl Isothiourea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Culturally Aware Adjuvant Endocrine Therapy (AET) Non-Initiation Intervention (Experimental): Participants will have two (2), 60 minute, individual sessions with a nurse practitioner via videoconferencing (in person or via telephone) and complete three (3) questionnaires at the time of enrollment, 1-month post-baseline, and 3-months post-baseline.
  Interventions: Behavioral: Culturally Aware Adjuvant Endocrine Therapy (AET) Non-Initiation Intervention

INTERVENTIONS:
Behavioral: Culturally Aware Adjuvant Endocrine Therapy (AET) Non-Initiation Intervention — One-to-One virtual (videoconference) behavioral intervention.

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of a brief, nurse-led intervention to support breast cancer survivors who have delayed initiation of hormonal therapy or who have concerns about starting hormonal therapy.

DETAILED DESCRIPTION:
This is a single-arm pilot trial to examine the feasibility and acceptability of a patient-centered, evidence-based, culturally competent, nurse-led intervention to encourage breast cancer survivors who have not begun taking adjuvant endocrine therapy (AET) to initiate the medication.

The research study procedures include:

* screening for eligibility
* two individual study intervention sessions
* study assessment follow-up questionnaires

This research study involves two individual sessions with a nurse practitioner which will take place via videoconferencing sessions either in-person or via telephone. Participants will also complete three brief questionnaire packets over the 12-week course of the study.

It is expected that up to 35 people will take part in this research study. The investigators plan to enrich the study sample for patients of a racial and/or ethnic minority in order to ensure the generalizability of the study findings.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 21 or older
* Diagnosis of early-stage (Stage 0-IIIB), hormone receptor-positive breast cancer
* Recommended to start AET at least 3 weeks prior and not currently taking AET OR recommended to start AET in the future and reports hesitations to start AET as determined by a score of >/= 4 (range =0-10) when asked "How hesitant are you about starting your recommended hormonal therapy? (0=Not at all hesitant and 10 = Extremely hesitant)"
* Ability to read and respond in English or Spanish
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* For at least 10 participants, identify as a member of a racial or ethnic minority community per self-report

Exclusion Criteria:

* Uncontrolled psychosis, active suicidal ideation, psychiatric hospitalization within the past year
* Cognitive impairment that prohibits participation in the study
* Undergoing primary treatment for other cancer (i.e., advanced stage cancer)
* Participating in a clinical trial involving AET

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Program Feasibility | Up to 3 months/12 weeks
  Feasibility will be demonstrated by enrollment (>50% of eligible and approached patients will enroll), retention (>70% of enrolled participants will complete the two intervention sessions) and attendance (≥70% of participants completing at least one session).
Program Acceptability | Up to 3 months/12 weeks
  Acceptability will be demonstrated by >75% of participants reporting average satisfaction scores greater than the mid-point of the Client Satisfaction Questionnaire. The total score range is 3-12, with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Adjuvant endocrine therapy (AET) Initiation | Baseline (within 1-week of consent), 1-month, and 3-months post-baseline
  Following the intervention, participants will be more likely to have started their AET. AET initiation will be measured by self-reported questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Jacobs, PhD, Principal Investigator — Massachusetts General Hospital
Locations (11):
- United States (11):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at St Elizabeth's Medical Center, Brighton, Massachusetts
  - Emerson Hospital/MGH Cancer Center, Concord, Massachusetts
  - Mass General at North Shore Cancer Center, Danvers, Massachusetts
  - Dana-Farber Brigham Cancer Center - Foxborough, Foxborough, Massachusetts
  - Dana-Farber Cancer Institute - Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber Brigham Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Mass General at Newton Wellesley Hospital, Newton, Massachusetts
  - Dana-Farber Brigham Cancer Center with South Shore Hospital, Weymouth, Massachusetts
  - Dana-Farber/New Hampshire Onoclogy-Hematology, Londonderry, New Hampshire

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Post KE, Dunderdale L, Datta S, Gutierrez N, Varella L, Horick N, Traeger L, Greer JA, Moy B, Temel JS, Jacobs JM. Development and refinement of a nurse-led, culturally sensitive intervention for adjuvant endocrine therapy initiation among patients with breast cancer. Eur J Oncol Nurs. 2025 Dec;79:103010. doi: 10.1016/j.ejon.2025.103010. Epub 2025 Oct 15. PMID 41172636